CLINICAL TRIAL: NCT04461353
Title: A Phase 1 Randomized Double Blind Placebo Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Orally Inhaled Aerosolized Hydroxychloroquine Sulfate in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Orally Inhaled Aerosolized Hydroxychloroquine Sulfate in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmoquine Therapeutics, Inc (Industry)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUL-01
Record Dates: First submitted 2020-06-23; First posted 2020-07-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-08

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: coronavirus; COVID-19; Hydroxychloroquine Sulfate; Hydroxychloroquine
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind placebo-controlled Phase 1 single-dose dose-escalation study to assess the safety, tolerability and PK of oral inhalation of AHCQ in healthy participants.
  A sentinel dose strategy will be employed and the decision to escalate to the next dose level, or deescalate or stop the study, will be based on review and analysis of all available blinded safety and tolerability data by the Safety Review Committee (SRC), which will make a recommendation to the Sponsor and the Sponsor will inform the PI of the recommendation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine Sulfate (Active Comparator): The study drug AHCQ will be administered by inhalation through the mouth. The starting dose will be 20 mg (Cohort A1) with a proposed subsequent dose of 50 mg (Cohort A2). At each dose level 8 participants (including at least 3 female participants and 3 participants older than 50 years old) will be enrolled. Six participants will receive the active study drug and 2 participants will receive placebo.
  Interventions: Drug: Aerolized Hydroxychloroquine Sulfate
- Placebo (Placebo Comparator): Placebo will be administered by inhalation through the mouth. It will be administered in both Cohort A1 and Cohort A2. Six participants will receive the active study drug and 2 participants will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aerolized Hydroxychloroquine Sulfate — sterile AHCQ 100 mg/mL for inhalation, is a clear solution packaged in clear glass vials and stored at room temperature.
  Other Names: AHCQ
  Arms: Hydroxychloroquine Sulfate
Other: Placebo — The placebo product and diluent solution is sodium chloride inhalation solution, United States Pharmacopeia (USP) 0.9%.
  Arms: Placebo

SUMMARY:
This study is 'A Randomized Phase 1 Double Blind Placebo Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Orally Inhaled Aerosolized Hydroxychloroquine Sulfate in Healthy Adult Volunteers.' The primary objectives are as follows:

* To assess the safety and tolerability of AHCQ administered as a single dose by oral inhalation in healthy individuals at escalating doses until either the maximum tolerated dose (MTD) is identified or 1 mL of a 50 mg/mL solution is administered.
* To determine the recommended Phase 2a dose (RP2D).

Secondary objectives:

• To characterize pharmacokinetics (PK) of single dose AHCQ in healthy individuals.

DETAILED DESCRIPTION:
Study Design:

This is a randomized, double-blind placebo-controlled Phase 1 single-dose dose-escalation study to assess the safety, tolerability and PK of oral inhalation of AHCQ in healthy participants.

Escalating single doses of AHCQ will be studied in healthy participants. The study drug will be administered by inhalation through the mouth, and participants will be encouraged to exhale through the nose. The study drug, AHCQ, will be administered starting at an initial dose of 20 mg (Cohort A1, 1 mL of 20 mg/mL AHCQ solution) with a proposed subsequent doses of 50 mg (Cohort A2, 1 mL of 50 mg/mL AHCQ).

Number of Participants (Planned):

Two dose levels are planned to be evaluated. Each cohort will comprise 8 participants (6 active, 2 placebo). Therefore, 16 participants will initially be planned to be enrolled in the study. Additional participants may be enrolled if one or more enrolled participants do not complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent.
2. Males or females aged ≥18 years old.
3. Good general health as determined by no acute illness and no clinically significant abnormal findings on medical history, vital signs, laboratory tests, or physical examination at screening that, in the opinion of the PI, would interfere with study drug administration, jeopardize the safety of the study participant, or impact the validity of the study results; participants with stable chronic illness are allowed at the discretion of the PI.
4. An interpretable 12-lead ECG with a corrected QT (QTc) interval ≤450 ms, according to Bazett's formula, without evidence of clinically significant abnormal findings.
5. Normal FEV1/FVC ratio, defined as any value above 0.7 or above the lower 5th percentile of normal AND FEV1 >80% of predicted or above the lower 5th percentile of normal.
6. Pulse oximetry 02 saturation ≥95% in room air.
7. Negative test result for COVID-19 within 7 days of Day 1 AND concurrent with local hospital policy:

   * A nasopharyngeal swab tested with the ID NOW COVID-19 assay (Abbot). OR
   * A negative RNA-based test result of an oropharyngeal or nasopharyngeal swab or saliva sample performed according to CLIA/CLEP.
8. Females of child-bearing potential must be non-pregnant, non-lactating, have a negative urine pregnancy test at screening, and agree to use an acceptable form of birth control for 200 days after the last administration of the study drug. Females are considered of non-childbearing potential if they are postmenopausal (last menstrual period at least 1 year before screening) or have been surgically sterilized (documented hysterectomy, tubal ligation, or bilateral oophorectomy) for at least 6 months at screening.
9. Willing to comply with protocol-defined procedures and complete all study visits.
10. Willing to use the Inhalation System and exhale through the nose.
11. Adequate venous access in the left or right arm to allow collection of required blood samples.
12. Participant understands and communicates in English.
13. Serum Potassium level ≥3.5 mEq/L, Serum Magnesium level ≥1.5 mg/dL, and Serum Calcium ≥8.5 mg/dL.

Exclusion Criteria:

1. Any self-reported symptoms of influenza-like or COVID-19-like illness in the 14 days preceding the study visit: Fever >101.4 °F, sore throat, nasal congestion, post-nasal discharge, shortness of breath, gastrointestinal distress, wheezing, cough, headache, or fatigue.
2. Any history of diagnosed chronic lung disease, including but not limited to asthma or chronic obstructive lung disease.
3. Symptoms of seasonal allergies or use of any drugs for seasonal allergies or any inhaled (oral/nasal) drugs in the 2 weeks prior to Day 1. Mild seasonal allergy symptoms that have not altered sleep or activity patterns nor required use of over-the-counter (OTC) or prescription medications are allowed.
4. Any close contact exposure in the past 28 days to a person who was diagnosed as having COVID-19, with or without laboratory confirmation, during that close contact exposure or in the ensuing 14 days OR a similar encounter with a person who was determined to have suspected COVID-19, defined by that person being ordered to enter isolation for that indication by a medical authority. Close contact is defined as being within approximately 6 feet of a COVID-19 case for a prolonged (>10 minutes) period of time and can occur while caring for, living with, visiting, or sharing a healthcare waiting area or room with a COVID-19 patient OR having direct contact with infectious secretions of a COVID-19 patient (e.g., being coughed on), if such contact occurred while not wearing the recommended personal protective equipment for that type of contact [e.g., gowns, gloves, N95 respirator (or equivalent), eye protection].
5. Any participant with a history of SARS-CoV-2 infection that was confirmed by testing or diagnosed without testing within 4 weeks preceding Day 1. If infection occurred more than 4 weeks prior, candidates may be enrolled if they meet the rest of the eligibility criteria.
6. Any participant with a history severe respiratory illness that required hospitalization in the 60 days preceding Day 1 OR any participant with a history severe respiratory illness that required hospitalization in the preceding 120 days without full recovery.
7. Participation in another clinical study that involved treatment with an investigational product or device within 30 days of screening or during the study.
8. Participants with a known history of human immunodeficiency virus (HIV) infection.
9. Known, active hepatitis A, B, or C infection.
10. History of bronchospasm in response to use of an inhalation device.
11. Use of any prescription medication (except oral contraceptives) during the 30 days prior to study dosing that may affect drug absorption, metabolism and excretion, prolong the QTc interval, affect drug efficacy, or increase the risk of adverse reactions, unless approved by the Principal Investigator.
12. Use of any OTC product, herbal product, diet aid, hormone supplement, etc., within 7 days prior to dosing unless approved by the Principal Investigator.
13. Unwilling or unable to provide written informed consent.
14. Any known hypersensitivity to quinolines (e.g., hydroxychloroquine, chloroquine, primaquine, quinine) or known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency or any contraindication to oral hydroxychloroquine.
15. Known retinopathy, fundus disease, or macular disease.
16. Diagnosis of long QT Syndrome.
17. Smoking of tobacco or non-tobacco substances, or vaping, within the last 6 months.
18. Severe obesity (body mass index [BMI] ≥35 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Incidences of treatment-emergent adverse events (TEAEs) as assessed by TGSHAAV (September 2007) or CTCAE version 5.0 | after treatment (Day 1) through to Day 30
  TEAEs (defined as AEs with onset after study drug administration or existing AEs that worsen in severity after study drug administration)
Change from baseline in clinical laboratory test results for CBC with differential | Screening and Day 8
  Blood sample collected for CBC with differential will be assessed from baseline (at screening)
Incidence of abnormal laboratory test results for CBC with differential at Screening | Screening
  Screening blood sample collected for CBC with differential, counting the number of abnormal clinical tests
Incidence of abnormal laboratory test results for CBC with differential - Day 8 | Day 8
  Day 8 blood sample collected for CBC with differential
Changes from baseline for blood glucose | Screening and Day 1
  Blood sample collected for blood glucose and measured with a glucometer
Incidence of abnormal laboratory test results for chemistry -Screening | Screening
  Blood sample collected for chemistry panel (albumin, total protein, ALP, ALT, AST, direct and indirect bilirubin, GGT, BUN, creatinine, glucose, bicarbonate, calcium, chloride, magnesium, phosphate, potassium, sodium, and LDH)
Incidence of abnormal laboratory tests results for chemistry - Day 8 | Day 8
  Blood sample collected for chemistry panel (albumin, total protein, ALP, ALT, AST, direct and indirect bilirubin, GGT, BUN, creatinine, glucose, bicarbonate, calcium, chloride, magnesium, phosphate, potassium, sodium, and LDH)
Incidence of abnormal laboratory tests results for urinalysis - Screening | Screening
  Collection of urine sample to test pH, specific gravity, protein, glucose, ketones, urobilinogen, bilirubin, leukocyte esterase, squamous cells, epithelial cells, clarity, bacteria, blood
Incidence of abnormal laboratory tests results for urinalysis- Day 8 | Day 8
  Collection of urine sample to test pH, specific gravity, protein, glucose, ketones, urobilinogen, bilirubin, leukocyte esterase, squamous cells, epithelial cells, clarity, bacteria, blood
Changes in vital signs from baseline (pre-dose) - respiratory rate | Screening, Day 1, Day 2 and Day 8
  The Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials (September 2007) (TGSHAAV) will be used as the primary criteria for assessment of clinical abnormalities. Mild (17-20 breaths per minute) to Potentially Life Threatening (intubation)
Changes in vital signs from baseline (pre-dose)- temperature | Screening, Day 1, Day 2 and Day 8
  Oral temperature
Changes in vital signs from baseline (pre-dose) - seated blood pressure | Screening, Day 1, Day 2 and Day 8
  Systolic and diastolic blood pressure
Changes in vital signs from baseline (pre-dose) - pulse | Screening, Day 1, Day 2 and Day 8
  Heart rate measure by radial pulse rate (beats/min)
Changes in vital signs from baseline (pre-dose) - O2 saturation | Screening, Day 1, Day 2 and Day 8
  O2 saturation (%), measured by pulse oximeter. Graded as per TGSHAAV (September 2007) from Moderate (pulse oximeter <92%) to Potentially Life Threatening (Life-threatening airway compromise; urgent intervention indicated)
Incidence of abnormal and physical examinations findings during Screening- general appearance | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - general appearance | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2- general appearance | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- general appearance | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening- neurological | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1- neurological | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2- neurological | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- neurological | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening - heart/cardiovascular | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - heart/cardiovascular | Day 1 (pre-dose, within 3 hours of dose)
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2 - heart/cardiovascular | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8 - heart/cardiovascular | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening - lungs | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - lungs | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2 - lungs | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8 - lungs | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening- abdomen | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - abdomen | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2- abdomen | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- abdomen | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during screening- endocrine | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - endocrine | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2- endocrine | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- endocrine | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening- extremities | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1- extremities | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2- extremities | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- extremities | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during Screening- lymphatic | Screening
  Physical exam by clinician. A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1- lymphatic | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2 - lymphatic | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8- lymphatic | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings during screening - skin | Screening
  A directed physical examination will be conducted
Incidence of abnormal and physical examinations findings on Day 1 - skin | Day 1
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 2 - skin | Day 2
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Incidence of abnormal and physical examinations findings on Day 8 - skin | Day 8
  Physical exam by clinician. A directed physical examination assessing and documenting changes from the previous visit, including any new abnormalities, will be conducted
Changes from baseline for pulmonary function tests (PFTs) - FEV1 | Screening, Day 1 at pre-dose (within 25 minutes of dose) and at +15 minutes, +1, +3 and +6 hours after study treatment, and on Day 2 and Day 8.
  Pulmonary function testing and recording of FEV1, both actual and percent predicted
Changes from baseline for pulmonary function tests (PFTs) - FVC | Screening, Day 1 at pre-dose (within 25 minutes of dose) and at +15 minutes, +1, +3 and +6 hours after study treatment, and on Day 2 and Day 8.
  Pulmonary function testing and recording of FVC, , both actual and percent predicted
Changes from baseline for pulmonary function tests (PFTs) - FEV1/FVC | creening, Day 1 at pre-dose (within 25 minutes of dose) and at +15 minutes, +1, +3 and +6 hours after study treatment, and on Day 2 and Day 8.
  Pulmonary function testing and recording of FEV1/FVC
Changes from baseline for ECG readings - QT interval | Screening and on Day 1 pre-dose (within 3 hours of dose) and approximately +2 and +6 hours, and on Days 2 and 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QT Interval (msec) will be the assessment parameter.
Changes from baseline for ECG readings - QTcB Interval | Screening and on Day 1 pre-dose (within 3 hours of dose) and approximately +2 and +6 hours, and on Days 2 and 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QTcB interval (msec) will be the assessment parameter.
Changes from baseline for ECG readings - QRS duration | Screening and on Day 1 pre-dose (within 3 hours of dose) and approximately +2 and +6 hours, and on Days 2 and 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QRS duration (msec) will be the assessment parameter.
Changes from baseline for ECG readings - PR interval | Screening and on Day 1 pre-dose (within 3 hours of dose) and approximately +2 and +6 hours, and on Days 2 and 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG PR interval (msec) will be the assessment parameter.
Changes from baseline for ECG readings - heart rate | Screening and on Day 1 pre-dose (within 3 hours of dose) and approximately +2 and +6 hours, and on Days 2 and 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG heart rate (beats/min) will be the assessment parameter.
Incidence of abnormal ECG - Screening | Screening
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QT Interval will be the assessment parameter.
Incidence of abnormal ECG- Day 1 | Day 1 pre-dose (within 3 hours of dose) and +2 and +6 hours
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QT Interval will be the assessment parameter.
Incidence of abnormal ECG - Day 2 | Days 2
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QT Interval will be the assessment parameter.
Incidence of abnormal ECG - Day 8 | Days 8.
  The ECG will be performed after the participant is allowed to rest seated for at least 5 minutes, before transferring to the examination bed/table for the ECG. ECG will be performed before PFTs or blood drawing.
  ECG QT Interval will be the assessment parameter.

SECONDARY OUTCOMES:
HCQ concentration in whole blood versus time profiles | Day 1 pre-dose (time 0) and +2, +3, +5, and +15 minutes after dose, and also +1, +2, +4 and +6 hours post-dose completion. Day 2 (+24±4 hours post dose) and Day 8.
  Blood samples for PK analysis will be collected via indwelling catheter or via direct venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Ohad S Bentur, MD, MHA, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.